CLINICAL TRIAL: NCT02546596
Title: The Effect of Electro-hyperthermia in Preoperative Radiotherapy Followed by Delayed Operation for Locally Advanced Rectal Cancer: Phase II Single Institutional Study
Brief Title: The Effect of Electro-Hyperthermia in Preoperative Radiotherapy for Locally Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei Hyperthermia Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YURO-H1
Record Dates: First submitted 2015-09-06; First posted 2015-09-11 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer; Hyperthermia
MeSH Terms: conditions — Rectal Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electro-hyperthermia plus radiation (Experimental): External beam radiation 40 Gy with 20 fractions (4 weeks) Electro-hyperthermia twice a week, one hour for each session
  Interventions: Device: Electro-hyperthermia

INTERVENTIONS:
Device: Electro-hyperthermia — Addition of electro-hyperthermia to radiation

SUMMARY:
Preoperative radiotherapy in locally advanced rectal cancer increases the possibility of complete resection and anal sphincter preservation. However, a treatment period of from 5 to 6 weeks is an obstacle of proper surgical intervention. Also, radiotherapy itself is confronting challenges for maximizing the therapeutic effect and minimizing the side effects. Electro-hyperthermia is appropriate treatment method to solve these kinds of problems. In this clinical trial, therapeutic effect of the high-frequency electro-hyperthermia is to be verified during preoperative radiotherapy for locally advanced rectal cancer. The ultimate goal is to establish a safe and effective treatment protocol.

DETAILED DESCRIPTION:
Preoperative radiotherapy in locally advanced rectal cancer increases the possibility of complete resection and anal sphincter preservation. However, a treatment period of from 5 to 6 weeks is an obstacle of proper surgical intervention. Also, radiotherapy itself is confronting challenges for maximizing the therapeutic effect and minimizing the side effects. Electro-hyperthermia is appropriate treatment method to solve these kinds of problems. In this clinical trial, therapeutic effect of the high-frequency electro-hyperthermia is to be verified during preoperative radiotherapy for locally advanced rectal cancer. The endpoint of the trial is treatment safety and non-inferiority of tumor regression to conventional schedule of preoperative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven rectal adenocarcinoma within 15 cm from anal verge
* Clinically T3-4 stage or positive lymph nodes
* Performance status 0-2
* Proper function of bone marrow, kidney, and liver

Exclusion Criteria:

* Past disease history of rectum
* Hereditary colorectal cancer
* Chronic inflammatory bowel disease
* Bower stenosis
* Active infection
* Myocardial infarction, uncontrolled arrhythmia, angina pectoris, or cardiac insufficiency within 6 months
* Pregnancy, nursing
* Unresected contemporary colon cancer
* Thermal hypersensitivity
* Too much subcutaneous fat in the abdominal and pelvic area

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
T stage (0 - 4), N (0 - 3) stage, tumor regression grade (0 - 4) | 3 months after curative surgery by surgical pathology report
  surgical pathology report

SECONDARY OUTCOMES:
Treatment toxicity (grade 0 - 5) | 5 years after curative surgery by clinical assessments
  clinical assessments

CONTACTS AND LOCATIONS:
Overall Officials: Sei Hwan You, MD, Study Director — Yonsei Hyperthermia Study Group
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Derived] Lee Y, Kim S, Cha H, Han JH, Choi HJ, Go E, You SH. Long-Term Feasibility of 13.56 MHz Modulated Electro-Hyperthermia-Based Preoperative Thermoradiochemotherapy in Locally Advanced Rectal Cancer. Cancers (Basel). 2022 Mar 1;14(5):1271. doi: 10.3390/cancers14051271. PMID 35267579